CLINICAL TRIAL: NCT06991257
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF AN ORAL BRANCHED-CHAIN KETOACID DEHYDROGENASE KINASE INHIBITOR, PF-07328948, IN ADULTS WITH HEART FAILURE (BRANCH-HF)
Brief Title: A Study to Learn About the Study Medicine Called PF-07328948 in Adults With Heart Failure (BRANCH-HF)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4921003; 2024-518438-94-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure with mildly reduced ejection; Heart Failure with preserved ejection fraction
MeSH Terms: conditions — Heart Failure | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ARM 1 (Placebo Comparator): Placebo Participants will receive Placebo for up to 36 weeks
  Interventions: Drug: Placebo
- ARM 2 (Experimental): Low dose PF-07328948 Participants will receive PF-07328948 for up to 36 weeks
  Interventions: Drug: Low Dose PF-07328948
- ARM 3 (Experimental): Medium dose PF-07328948 Participants will receive PF-07328948 for up to 36 weeks
  Interventions: Drug: Medium Dose PF-07328948
- ARM 4 (Experimental): High dose PF-07328948 Participants will receive PF-07328948 for up to 36 weeks
  Interventions: Drug: High Dose PF-07328948

INTERVENTIONS:
Drug: Placebo — ARM 1
  Arms: ARM 1
Drug: Low Dose PF-07328948 — ARM 2
  Other Names: low dose
  Arms: ARM 2
Drug: Medium Dose PF-07328948 — ARM 3
  Other Names: medium dose
  Arms: ARM 3
Drug: High Dose PF-07328948 — ARM 4
  Other Names: High dose
  Arms: ARM 4

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (PF-07328948) for the possible treatment of heart failure (HF).

DETAILED DESCRIPTION:
All participants in this study will take either the study medicine (PF-07328948) tablets, or placebo tablets, once daily, by mouth, every day for 36 weeks. The study determines if the study medicine (PF-07328948) is safe and effective compared to placebo in people with heart failure who are already taking standard-of-care medications for heart failure that include sodium-glucose cotransporter 2 (SGLT2) inhibitors. Participants will be involved in this study for about 48 weeks. During this time, participants will visit the study clinic 15 times. In general, 5 of these visits may be performed at home by phone and the other 10 visits will take place at the study site.

ELIGIBILITY:
This study is seeking participants who are:

Key Inclusion Criteria include:

* aged 18 years to < 80 years
* clinically confirmed to have a diagnosis of heart failure for at least 3 months
* New York Heart Association Class II-IV symptoms
* left ventricular ejection fraction greater than 40%
* Kansas City Cardiomyopathy Questionnaire-23 Total Symptom Score < 85
* Six-minute walking distance greater than 75 meters

Key Exclusion Criteria include:

* Type 1 diabetes mellitus, liver cirrhosis or any condition that can possibly affect how the medicine is absorbed into the body.
* Major surgery scheduled for the duration of the study, affecting walking ability in the opinion of the study doctor.
* History of heart transplantation, or currently listed for a heart transplant, or current planned use of IV vasodilators and/ or inotropes
* Prior intolerance/known hypersensitivity to an SGLT2 inhibitor or contraindication to an SGLT2 inhibitor

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-11-16 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Clinical Events | over 36 weeks
  Adjudicated cardiovascular death and worsening heart failure events through 36 weeks.
Change From Baseline in 6-Minute Walk Test (6MWD) | Baseline, week 36 post-dose
  A submaximal exercise test that measures the distance the participant can walk within prescribed time of 6 minutes. Participants are asked to perform the test at a pace comfortable to them with as many breaks as needed. The total distance walked is recorded.
Change From Baseline in Kansas City Cardiomyopathy Questionnaire Overall Total Symptom Score (KCCQ-23 TSS) | Baseline, week 36
  KCCQ is a 23-item heart-failure specific questionnaire quantified into the following scores: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life, and self-efficacy, total symptom score, overall summary score, and clinical summary score. To facilitate interpretation, all scores are presented on a scale of 0 to 100 points, with lower scores indicating more severe symptoms and/or limitations, and a score of 100 indicating no symptoms, no limitations, and excellent quality of life.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Baseline, up to week 40
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE that, at any dose, results in 1 or more of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 40 that were absent before treatment or that worsened relative to pre-treatment state. AEs include both serious and non-serious adverse events.
Change From Baseline in Kansas City Cardiomyopathy Questionnaire Overall Symptom Score (KCCQ-23 TSS) and physical limitation in participants taking PF-07328948 vs. placebo on HF disease-specific health status related to HFmrEF/HFpEF. | Baseline, week 36
  KCCQ is a 23-item participant-completed questionnaire that assesses health status and health-related quality of life in participants with heart failure. Eight domain scores were calculated for the KCCQ: Physical limitation, Social limitation, Quality of life, Self-efficacy, Symptom stability, Symptom frequency, Symptom burden, and Total symptoms (calculated as the mean of Symptom frequency and Symptom burden scores). Two summary scores are also calculated: Clinical Summary (calculated as mean of Physical limitation and Total symptom scores) and Overall Summary (calculated as mean of Physical limitation, Social limitation, Total symptoms, and Quality of life scores). Domain and summary scores were scaled to range from 0 (minimum) to 100 (maximum); higher scores represent better health status.
Change From Baseline in 6-minute walk test distance (6MWD) in participants taking PF-07328948 vs. placebo on HF disease-specific health status related to HFmrEF/HFpEF. | Baseline, week 36
  A submaximal exercise test that measures the distance the participant can walk within prescribed time of 6 minutes. Participants are asked to perform the test at a pace comfortable to them with as many breaks as needed. The total distance walked is recorded.
CPET Substudy) : Change From Baseline in Peak Oxygen Consumption (pVO2) at Week 36 | Baseline, Week 36
  Cardiopulmonary exercise testing
Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration at Week 36 | Baseline, Week 36
  NT-proBNP is a biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ LV wall stress).
Change From Baseline in Kansas City Cardiomyopathy Questionnaire Overall clinical symptom Score (KCCQ-23 CSS) and physical limitation) in participants taking PF-07328948 vs. placebo on HF disease-specific health status related to HFmrEF/HFpEF. | Baseline, week 36
  KCCQ is a 23-item participant-completed questionnaire that assesses health status and health-related quality of life in participants with heart failure. Eight domain scores were calculated for the KCCQ: Physical limitation, Social limitation, Quality of life, Self-efficacy, Symptom stability, Symptom frequency, Symptom burden, and Total symptoms (calculated as the mean of Symptom frequency and Symptom burden scores). Two summary scores are also calculated: Clinical Summary (calculated as mean of Physical limitation and Total symptom scores) and Overall Summary (calculated as mean of Physical limitation, social limitation, Total symptoms, and Quality of life scores). Domain and summary scores were scaled to range from 0 (minimum) to 100 (maximum); higher scores represent better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (20):
  - National Heart Institute, Beverly Hills, California
  - Orange County Research Center, Lake Forest, California
  - Comprehensive Cardiovascular Care, Santa Maria, California
  - FOMAT Medical Research, Santa Maria, California
  - FWD Clinical Research, Boca Raton, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Infinite Clinical Research, Miami, Florida
  - Flourish Research Acquisition, LLC dba Flourish Research - North Miami, Miami, Florida
  - Amavita Research Services, North Miami Beach, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Chicago Medical Research, Hazel Crest, Illinois
  - NexGen Research, Fort Wayne, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Velocity Clinical Research, Lincoln, Pioneer Heart Institute, Lincoln, Nebraska
  - NexGen Research, Lima, Ohio
  - Headlands Horizons, LLC dba Headlands Research-Brownsville, Brownsville, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Northwest Houston Heart Center, Tomball, Texas
- Bulgaria (9):
  - Diagnostic Consultative Center - 1 Lom EOOD, Lom, Montana
  - Diagnostic Consultative Center "Ascendent", Sofia, Sofia (stolitsa)
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia (stolitsa)
  - "Multiprofile Hospital for Active Treatment Puls" AD, Blagoevgrad
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova AD, Gabrovo
  - Medical Center Hera - Kyustendil EOOD, Kyustendil
  - MHAT - Heart and Brain, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - MHAT Hadzhi Dimitar, Sliven
- Canada (14):
  - Richmond Clinical Trials, Richmond, British Columbia
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - ACV Clinic, Greater Sudbury, Ontario
  - CardioQuest Research Centre, Sarnia, Ontario
  - Corcare, Toronto, Ontario
  - Community Care Building, Winchester, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - CHU de Quebec - Université Laval - Hotel Dieu de Quebec, Québec, Quebec
  - Clinique de Médecins Spécialistes, Shebrooke, Quebec
  - Diex Recherche Sherbrooke Est, Sherbrooke, Quebec
  - Centre intégré de santé et de services sociaux de Lanaudière - Hopital Pierre-Le Gardeur., Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
- Czechia (5):
  - Sdružené Zdravotnické Zařízení Krnov, Krnov, Moravskoslezský kraj
  - Kardiologicka ambulance Brno s.r.o., Brno-Královo Pole
  - EFERTUS healthcare s.r.o., Brno-Židenice
  - EDUMED s.r.o., Jaroměř
  - VASOMED Clinic s.r.o., Ostrava
- France (3):
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain, Loire-atlantique
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, Provence-Alpes-Côte d'Azur Region
  - Chu Grenoble Alpes, Grenoble
- Hungary (6):
  - Da Vinci Magánklinika, Pécs, Baranya
  - CMed Rehabilitacios es Diagnosztikai Kozpont, Székesfehérvár, Fejér
  - Ezüstfény Klinika Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Jahn Ferenc Dél-pesti Hospital, Budapest
  - New Medical Center Kft., Sopron
- Japan (20):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Nagoya Tokushukai General Hospital, Kasugai, Aichi-ken
  - Seikeikai New Tokyo Heart Clinic, Matsudo, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Koga General Hospital, Koga, Ibaraki
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - National Hospital Organization Mie Chuo Medical Center, Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - National Hospital Organization Saitama Hospital, Wako, Saitama
  - Tokyo Metropolitan Toshima Hospital, Itabashi-ku, Tokyo
  - Showa General Hospital, Kodaira-shi, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - NewHeart Watanabe Institute, Suginami, Tokyo
  - Sekino Hospital, Toshimaku, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi
  - Nagasaki Harbor Medical Center, Nagasaki
- Poland (4):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - SP ZOZ w Puławach, Puławy, Lublin Voivodeship
  - NZOZ Sopockie Centrum Badan Kardiologicznych Pro Cordis Pawel Miekus, Sopot, Pomeranian Voivodeship
  - Kardio Brynow, Katowice, Silesian Voivodeship
- Research and Cardiovascular Corp., Ponce, Puerto Rico
- Spain (8):
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (5):
  - Ninewells Hospital and Medical School, Dundee, Dundee CITY
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - St Richard's Hospital, Chichester, WEST Sussex
  - South Eastern Health and Social Care Trust, Belfast
  - Wycombe General Hospital, High Wycombe

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921003